CLINICAL TRIAL: NCT00198094
Title: A Randomized Double-Blind Comparison of Sertraline With Early Alprazolam XR Co-Administration vs Sertraline/Placebo for Primary Care Panic Disorder Patients
Brief Title: A Study of Sertraline and Early Alprazolam XR Administration Versus Sertraline Only in Panic Disorder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Pfizer (Industry); University of Pennsylvania (Other); University of South Florida (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0311-34; IU 1003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sertraline and Alprazolam XR

SUMMARY:
The primary objective for the study is to test the hypothesis that sertraline plus alprazolam XR will result in superior early stabilization of primary care PD patients versus sertraline/placebo over a 12-week treatment period. The secondary objectives of the study are a) to assess withdrawal symptoms during alprazolam XR taper (weeks 5-7 of the 12-week trial) and after discontinuation, b) to compare physical health outcomes, medical services utilization, and cost-effectiveness of the two study interventions across the 12-week treatment period and subsequent three month maintenance treatment with sertraline alone, and c) to assess whether early co-administration of sertraline/ alprazolam XR will result in greater maintenance of treatment response than sertraline/placebo over the three months following the 12 week acute treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include men and women over the age of eighteen;
* the ability to give written informed consent;
* current principal or co-principal psychiatric diagnosis of panic disorder with or without agoraphobia based on DSM-IV criteria (American Psychiatric Association, 1994);
* willing to use an effective means of contraception;
* free of psychoactive medications for at least 2 weeks prior to study enrollment;
* not actively be suicidal.

Exclusion Criteria:

* actively suicidal;
* medical conditions for which either sertraline or alprazolam XR would be contraindicated;
* recent six month history of substance or alcohol abuse;
* history or presence of psychotic or bipolar disorder;
* women who are pregnant or breastfeeding;
* history or presence of a seizure disorder or a known history of more than one childhood febrile seizure;
* presence of a personality disorder severe enough to compromise the investigator's ability to evaluate the efficacy and safety of the study medication;
* concomitant therapy with other psychotropic medication(s);
* clinically significant abnormality during physical examination, vital signs, EKG, urine drug screen, or laboratory tests at the screen visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Panic symptoms scale score
CGI-I
CGI-S

SECONDARY OUTCOMES:
Sheehan Disability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Goddard, M.D., Principal Investigator — Indiana University; Karl Rickles, M.D., Principal Investigator — University of Pennsylvania; David Sheehan, M.D., M.B.A., Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - University of South Florida, Department of Psychiatry and Behavioral Medicine, Tampa, Florida
  - University Hospital Outpatient Center, Psychiatry, Indianapolis, Indiana
  - University of Pennsylvania, Mood and Anxiety Disorders Section, Philadelphia, Pennsylvania

REFERENCES:
- [Result] A randomized double-blind comparison of sertraline with early alprazolam XR Co-administration vs. sertraline/placebo for panic disorder. Goddard AW, Ball SG, Hastings AK, Shekhar A, Rickels K, Rynn M, Janavs J, Sheehan DV. BIOLOGICAL PSYCHIATRY 57 (8): 62S-62S 220 Suppl. S, APR 15 2005. IDS Number: 915VE ISSN: 0006-3223